CLINICAL TRIAL: NCT03881748
Title: A Randomized Phase II Pilot Clinical Trial of Acupuncture for Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Clinical Trial of Acupuncture for Chemotherapy-Induced Peripheral Neuropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staff
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE4Y18
Record Dates: First submitted 2019-03-18; First posted 2019-03-19 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Peripheral Neuropathy
Keywords: Acupuncture
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: 1) manual acupuncture twice a week for 20 treatments or 2) electro-acupuncture twice a week for 20 treatments. Multiple assessments will be performed at baseline and approximately every 2 weeks for a total of 16 weeks while subjects are on study.
Who Masked: Care Provider
Masking Description: A research assistant blind to group assignment will distribute and collect the results of the FACT/GOG-Ntx subscale, FACT-G, TNSc, NPS, QST, GPT, Unipedal Stance balance test, and medication use per the study calendar. In addition, data about the subject's past medical history including cancer details and relevant medical conditions (e.g., diabetes mellitus and peripheral vascular disease) will be collected. This data will not be seen by the acupuncturists while the subject is receiving treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual acupuncture (Experimental): Insertion of very thin, solid, sterile, stainless steel needles into the skin at specific points.
  Interventions: Other: Manual acupuncture
- Electro-acupuncture (Experimental): Insertion of very thin, solid, sterile, stainless steel needles into the skin at specific points with additional application of weak electrical stimulation
  Interventions: Other: Electro-acupuncture

INTERVENTIONS:
Other: Manual acupuncture — Manual acupuncture twice a week for 20 treatments.
  Acupuncture will be administered on an outpatient basis in private rooms with participants lying supine. The acupuncturist will disinfect the selected acupuncture points with alcohol and then needle them so that the participant achieves a "de qi" sensation if possible, which is often described as a pressure or achiness feeling. Acupuncture needles will be left in place for approximately 20 minutes.
  Arms: Manual acupuncture
Other: Electro-acupuncture — Electro-acupuncture twice a week for 20 treatments.
  Acupuncture will be administered on an outpatient basis in private rooms with participants lying supine. The acupuncturist will disinfect the selected acupuncture points with alcohol and then needle them so that the participant achieves a "de qi" sensation if possible, which is often described as a pressure or achiness feeling. Acupuncture needles will be left in place for approximately 20 minutes.
  Electrical stimulation will be applied to the needles concomitantly and continuously to acupuncture points by placing lead wires on the needles connected to an electro-acupuncture stimulator such as the Model IC-1107. The stimulator will be set on the Dense-Disperse wave setting with low frequency at 2-10 Hz and high frequency at 100-110 Hz. The needles will not be manually stimulated after electrical stimulation is applied.
  Arms: Electro-acupuncture

SUMMARY:
The goal of this clinical research study is to learn if one acupuncture treatment approach is more effective than another in helping to relieve chemo-therapy induced neuropathy in cancer patients. If eligible to take part in this study, participants will be randomly assigned to 1 of 2 groups - group 1 participants will receive traditional acupuncture treatments 2 times a week for a total of 20 sessions. Group 2 participants will have acupuncture sessions with electrical stimulation 2 times a week for a total of 20 sessions.

DETAILED DESCRIPTION:
Peripheral neuropathy is a common problem among cancer patients who have received chemotherapy treatment. Peripheral neuropathy often causes weakness, numbness and pain, usually in the hands and feet. It can also affect other areas of the body. People with peripheral neuropathy generally describe the pain as stabbing, burning or tingling.

Acupuncture is a technique that may treat symptoms by inserting very thin, solid, sterile, stainless steel needles into the skin at specific points. Research has shown that acupuncture can reduce symptoms of pain and nausea by altering pain signaling along nerves. The effect of acupuncture can be enhanced by additional movement of the needles called manual acupuncture, which involves rotating the needle and moving it up and down. Another type of acupuncture is called electro-acupuncture, which involves running a low level electrical current between two needle points. Preliminary studies indicate that acupuncture may also be helpful to treat chemotherapy related neuropathy. This trial will determine the relative effects of both manual acupuncture and electro-acupuncture for treating chronic chemotherapy-induced neuropathy.

Participants will be assigned to one of two groups: 1) manual acupuncture twice a week for 20 treatments or 2) electro-acupuncture twice a week for 20 treatments. Multiple assessments will be performed at baseline and approximately every 2 weeks for a total of 16 weeks while subjects are on study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have the ability to understand English, sign a written informed consent document, and be willing to follow protocol requirements.
* History of a diagnosis of cancer, verifiable through documentation in a medical record.
* Participants must have neuropathy ≥1 according to CTCAE v 4.0 scale or a neuropathy score of >3 on a 0-10 scale despite previous treatment, which may include Neurontin, Cymbalta and/or Lyrica.
* The participant's previous chemotherapy treatment must have included a taxane (paclitaxel, nab-paclitaxel, or docetaxel) or platinum (cisplatin, oxaliplatin, or carboplatin) and considered the primary cause of the neuropathy by the medical team.
* More than 6 months since last treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* Willingness to comply with all study interventions of acupuncture and follow-up assessments.

Exclusion Criteria:

* Current active treatment with chemotherapy, radiation or surgery in the past 3 months or planned treatment during this study protocol period. Hormonal therapy is allowed.
* Treatment with any neuropathic agent including taxane, platinum, vinca alkaloid, or bortezomib chemotherapy within the past 6 months.
* Local infection at or near the acupuncture site. (Although acupuncture is a minimally invasive procedure, participants will be excluded if there is an indication of infection.)
* Physical deformities that could interfere with accurate acupuncture point location.
* Concurrent use of other alternative medicines such as herbal agents and high dose vitamins and minerals.
* Known coagulopathy or taking heparin (including low molecular weight heparin) at full anti-coagulation doses (prophylaxis is allowed) or Coumadin at any dose. Participants on aspirin or non-steroidal anti-inflammatories or other antiplatelet medicines will be allowed to participate.
* Platelets < 50 H K/UL in the past 30 days.
* White Blood Cells (WBCs) < 3.0 K/UL or absolute neutrophil count (ANC) <1,500 K/UL) in the past 30 days.
* Active Central Nervous System (CNS) disease. (The action for acupuncture may be associated with central nervous system activity, and participants with CNS pathology may respond differently to treatment than the general population.)
* Implanted electrical device such as cardiac pacemaker, insulin pump, or pain pump.
* Mental incapacitation or significant emotional or psychological disorder that, in the opinion of the investigators, precludes study entry. (These participants may not be able to cooperate with this slightly invasive procedure or with the data collection process.)
* Currently pregnant. (Certain acupuncture applications have been reported to stimulate uterine contractions.)
* History of diabetic neuropathy, neuropathy related to HIV, or other medical causes of chronic neuropathy in the baseline assessment including past medical history, any history of diabetes, alcoholism, and vitamin B.
* Previous acupuncture treatment for any indication within 30 days of enrollment.
* Planned or actual changes in type of medications that could affect symptoms related to chemotherapy-induced peripheral neuropathy (CIPN). New medications for the treatment of CIPN are not allowed during the study. Subjects need to be on stable doses of CIPN medications for 4 weeks.
* Grade III lymphedema or lymphedema considered severe by the treating clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Treatment completion rate | Up to 12 weeks from start of study.
  Percent of participants that complete the treatment protocol, with completions being defined as receiving at least 20 acupuncture treatments within 2 weeks of the scheduled course of treatments (Which is 12 weeks).

SECONDARY OUTCOMES:
Cancer-specific, health-related quality of life as measured by FACT-G | At 2, 4, 6, 8, 10, and 14 weeks after start of treatment.
  Cancer-specific, health-related quality of life as measured by Functional Assessment of Cancer Therapy: General (FACT-G) questionnaire. The range of scores lies on a spectrum of 0 - 108, with higher scores indicating better quality of life.
Peripheral neuropathy or neuropathy as measured by (Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity subscale (FACT/GOG-Ntx) | At 2, 4, 6, 8, 10, and 14 weeks after start of treatment.
  The Ntx subscale is an 11-item questionnaire to assess neurotoxic effects of chemotherapy with scores ranging on a scale of 11-44.
Quality of life as measured by Total Neuropathy Score - Clinically Based (TNSc) | At 2, 4, 6, 8, 10, and 14 weeks after start of treatment.
  The Total Neuropathy Score - Clinically Based (TNSc) scale is a 10-item scale assessing chemotherapy-induced peripheral neuropathy with scores ranging on a scale of 0-44. Higher scores indicate worse symptoms.
Quality of life as measured by Neuropathy Pain Scale (NPS) | At 2, 4, 6, 8, 10, and 14 weeks after start of treatment.
  The Neuropathy Pain Scale (NPS) is a 10-item scale assessing neuropathic pain with scores ranging on a scale of 0-100. Higher scores indicate worse symptoms.
Change in participant's ability to detect thermal sensory stimuli as measured by Quantitative Sensory Testing (QST) | At 2, 4, 6, 8, 10, and 14 weeks after start of treatment.
  Threshold detection of thermal sensory stimuli as measured by Quantitative Sensory Testing (QST) to assess change in participant's ability to detect thermal sensory stimuli.
Change in participant's ability to detect vibration sensory stimuli as measured by Quantitative Sensory Testing (QST) | At 2, 4, 6, 8, 10, and 14 weeks after start of treatment.
  Threshold detection of vibration sensory stimuli as measured by Quantitative Sensory Testing (QST) to assess change in participant's ability to detect vibration sensory stimuli.
Change in hand function as measured by Grooved Pegboard Test (GPT) | At 2, 4, 6, 8, 10, and 14 weeks after start of treatment.
  Times the ability of subjects to complete insertion of 25 shaped pegs and is a surrogate for hand function. Subjects will be asked to complete the GPT twice and the time will be averaged for each assessment time point. An increasing time to complete the task would indicate worsening hand function due to neuropathy symptoms. Change in time taken to complete task will be reported.
Change in balance as measured by Unipedal Stance balance test | At 2, 4, 6, 8, 10, and 14 weeks after start of treatment.
  Participants will perform a unipedal stance with eyes open for a goal of 45 seconds and will be allowed a total of 3 trials to achieve the 45 seconds with the highest time recorded. A decreasing time of unipedal stance would indicate worsening balance due to neuropathy symptoms. Change in time will be reported.
Use of neuropathic and pain medications | At 2, 4, 6, 8, 10, and 14 weeks after start of treatment.
  Change in number of medications after treatment (decrease in medications being positive change). These medications may include NSAIDS, acetaminophen, opioid medications (e.g., morphine, oxycodone), amitriptyline, neurontin, pregabalin, carbamezapine, or other related medications.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States